CLINICAL TRIAL: NCT02076347
Title: Comparison of Two Pharmacist-led Population Management Approaches to Increase Monitoring of Vitamin B12 and Serum Creatinine Levels for Patients on Metformin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Kelli Barnes, Assistant Professor of Clinical Pharmacy, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2013H0307
Record Dates: First submitted 2014-02-26; First posted 2014-03-03 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2015-10

CONDITIONS: Type 2 Diabetes; Vitamin B12 Deficiency; Neuropathy; Anemia
Keywords: Metformin; Vitamin B12 Deficiency; Population Management; Pharmacist
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Vitamin B 12 Deficiency; Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Office visit-based intervention (Experimental)
  Interventions: Behavioral: Office visit intervention
- Electronic message-based intervention (Experimental)
  Interventions: Behavioral: Electronic Message Intervention

INTERVENTIONS:
Behavioral: Office visit intervention — Pharmacist communicates monitoring recommendations to physician through the electronic medical record prior to a scheduled patient office visit
  Arms: Office visit-based intervention
Behavioral: Electronic Message Intervention — Pharmacist communicates need for monitoring directly to patients and instructs them to obtain monitoring on their own time without need for an office visit with physician
  Arms: Electronic message-based intervention

SUMMARY:
The purpose of this project is to compare two pharmacist-led population management strategies designed to increase the rate of appropriate monitoring of vitamin B12 and serum creatinine for patients taking metformin.

ELIGIBILITY:
Inclusion Criteria:

* On Metformin for at least one year
* Activated patient portal for electronic messaging
* Patient of an attending physician at Ohio State General Internal Medicine
* No serum vitamin B12 and/or no serum creatinine measurement in the past year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 489 (Actual)
Dates: Start 2014-02; Primary Completion 2014-08 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Percentage of patients in each arm who obtain monitoring of vitamin B12 as recommended | 6 months

SECONDARY OUTCOMES:
Number of patients with newly identified vitamin B12 deficiency | 6 months
Percentage of patients with newly identified vitamin B12 deficiency who have prior evidence of anemia upon chart review | within 6 months
  When a patient's serum vitamin B12 level comes back and is low the chart will be reviewed immediately to determine this. This could happen anytime during the 6 month study period.
Percentage of patients with newly identified vitamin B12 deficiency who have prior evidence of neuropathy upon chart review | within 6 months
  When a patient's serum vitamin B12 level comes back and is low the chart will be reviewed immediately to determine if neuropathy is also listed as a medical problem. This could happen anytime during the 6 month study period.

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University General Internal Medicine, Columbus, Ohio, United States

REFERENCES:
- [Derived] Matthews DE, Beatty SJ, Grever GM, Lehman A, Barnes KD. Comparison of 2 Population Health Management Approaches to Increase Vitamin B12 Monitoring in Patients Taking Metformin. Ann Pharmacother. 2016 Oct;50(10):840-6. doi: 10.1177/1060028016655180. Epub 2016 Jun 20. PMID 27323792